CLINICAL TRIAL: NCT01217307
Title: Metabolic Modulation With Metformin to Reduce Heart Failure After Acute Myocardial Infarction: Glycometabolic Intervention as Adjunct to Primary Coronary Intervention in ST Elevation Myocardial Infarction (GIPS-III): a Randomized Controlled Trial.
Brief Title: Metformin to Reduce Heart Failure After Myocardial Infarction
Acronym: GIPS-III
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Chris Lexis, Drs., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIPS-III 2010B257
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-07

CONDITIONS: ST Elevation Myocardial Infarction (STEMI); Coronary Artery Disease; Heart Failure; Diabetes
Keywords: Metformin; ST elevation myocardial infarction (STEMI); Coronary artery disease; Heart failure; Diabetes
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease; Heart Failure; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): metformin 500mg twice daily during 4 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo twice daily during 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500mg twice daily during 4 months
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Placebo twice daily during 4 months
  Arms: Placebo

SUMMARY:
The investigators will evaluate the effect of metformin therapy during 4 months in non-diabetic patients following ST-elevation myocardial infarction on left ventricular ejection fraction as measured with cardiac magnetic resonance imaging, compared to placebo.

DETAILED DESCRIPTION:
In this trial, the investigators will evaluate the effect of metformin therapy following ST-elevation myocardial infarction (STEMI) in a total of 380 non-diabetic patients. This trial is a randomized, double blind, controlled trial. The intervention, which consist of metformin 500mg twice daily or placebo twice daily, will commence within three hours after the percutaneous coronary intervention, and will be continued for 4 months. The primary endpoint is the difference between the two intervention groups (metformin vs placebo) in left ventricular ejection fraction, as measured with magnetic resonance imaging after 4 months. The investigators hypothesize that metformin therapy results in a significantly higher ejection fraction in this population.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis acute MI defined by chest pain suggestive for myocardial ischemia for at least 30 minutes, the time from onset of the symptoms less than 12 hours before hospital admission, and an ECG recording with ST- segment elevation of more than 0.1 mV in 2 or more leads.
* Successful primary PCI (post-procedural TIMI 2/3);
* At least one stent sized ≥ 3.0 mm;
* Eligible for 3T CMR imaging;
* Verbal followed by written informed consent.

Exclusion Criteria:

* rescue PCI after thrombolytic therapy;
* need for emergency coronary artery bypass grafting;
* creatinin >177 μmol/L measured pre-PCI;
* Younger than 18 years;
* Mechanical ventilation;
* Diabetes;
* Prior myocardial infarction;
* Contra-indication to metformin (see safety);
* The existence of a life-threatening disease with a life-expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iwan CC van der Horst, MD, PhD, Principal Investigator — Thorax Centre, University Medical Centre Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Al Ali L, Groot HE, Assa S, Lipsic E, Hummel YM, van Veldhuisen DJ, Voors AA, van der Horst ICC, Lam CS, van der Harst P. Predictors of adverse diastolic remodeling in non-diabetic patients presenting with ST-elevation myocardial infarction. BMC Cardiovasc Disord. 2023 Jan 23;23(1):44. doi: 10.1186/s12872-023-03064-7. PMID 36690932
- [Derived] de Koning MLY, Westenbrink BD, Assa S, Garcia E, Connelly MA, van Veldhuisen DJ, Dullaart RPF, Lipsic E, van der Harst P. Association of Circulating Ketone Bodies With Functional Outcomes After ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2021 Oct 5;78(14):1421-1432. doi: 10.1016/j.jacc.2021.07.054. PMID 34593124
- [Derived] Hartman MHT, Prins JKB, Schurer RAJ, Lipsic E, Lexis CPH, van der Horst-Schrivers ANA, van Veldhuisen DJ, van der Horst ICC, van der Harst P. Two-year follow-up of 4 months metformin treatment vs. placebo in ST-elevation myocardial infarction: data from the GIPS-III RCT. Clin Res Cardiol. 2017 Dec;106(12):939-946. doi: 10.1007/s00392-017-1140-z. Epub 2017 Jul 28. PMID 28755285
- [Derived] Eppinga RN, Kofink D, Dullaart RP, Dalmeijer GW, Lipsic E, van Veldhuisen DJ, van der Horst IC, Asselbergs FW, van der Harst P. Effect of Metformin on Metabolites and Relation With Myocardial Infarct Size and Left Ventricular Ejection Fraction After Myocardial Infarction. Circ Cardiovasc Genet. 2017 Feb;10(1):e001564. doi: 10.1161/CIRCGENETICS.116.001564. PMID 28100626
- [Derived] Eppinga RN, Hartman MH, van Veldhuisen DJ, Lexis CP, Connelly MA, Lipsic E, van der Horst IC, van der Harst P, Dullaart RP. Effect of Metformin Treatment on Lipoprotein Subfractions in Non-Diabetic Patients with Acute Myocardial Infarction: A Glycometabolic Intervention as Adjunct to Primary Coronary Intervention in ST Elevation Myocardial Infarction (GIPS-III) Trial. PLoS One. 2016 Jan 25;11(1):e0145719. doi: 10.1371/journal.pone.0145719. eCollection 2016. PMID 26808474
- [Derived] Lexis CP, van der Horst-Schrivers AN, Lipsic E, Valente MA, Muller Kobold AC, de Boer RA, van Veldhuisen DJ, van der Harst P, van der Horst IC. The effect of metformin on cardiovascular risk profile in patients without diabetes presenting with acute myocardial infarction: data from the Glycometabolic Intervention as adjunct to Primary Coronary Intervention in ST Elevation Myocardial Infarction (GIPS-III) trial. BMJ Open Diabetes Res Care. 2015 Dec 11;3(1):e000090. doi: 10.1136/bmjdrc-2015-000090. eCollection 2015. PMID 26688733
- [Derived] Lexis CP, van der Horst IC, Lipsic E, Wieringa WG, de Boer RA, van den Heuvel AF, van der Werf HW, Schurer RA, Pundziute G, Tan ES, Nieuwland W, Willemsen HM, Dorhout B, Molmans BH, van der Horst-Schrivers AN, Wolffenbuttel BH, ter Horst GJ, van Rossum AC, Tijssen JG, Hillege HL, de Smet BJ, van der Harst P, van Veldhuisen DJ; GIPS-III Investigators. Effect of metformin on left ventricular function after acute myocardial infarction in patients without diabetes: the GIPS-III randomized clinical trial. JAMA. 2014 Apr 16;311(15):1526-35. doi: 10.1001/jama.2014.3315. PMID 24687169
- [Derived] Lexis CP, van der Horst IC, Lipsic E, van der Harst P, van der Horst-Schrivers AN, Wolffenbuttel BH, de Boer RA, van Rossum AC, van Veldhuisen DJ, de Smet BJ; GIPS-III Investigators. Metformin in non-diabetic patients presenting with ST elevation myocardial infarction: rationale and design of the glycometabolic intervention as adjunct to primary percutaneous intervention in ST elevation myocardial infarction (GIPS)-III trial. Cardiovasc Drugs Ther. 2012 Oct;26(5):417-26. doi: 10.1007/s10557-012-6413-1. PMID 22968678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 191 | 189
Completed | 191 | 188
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 191 | 189 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.8) | 58.8 (11.5) | 58.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 144 | 141 | 285

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Left Ventricular Ejection Fraction
Description: The primary efficacy parameter of the GIPS-III trial is LVEF measured by cardiac MRI 4 months after randomization, based on an intention-to-treat analysis. It is hypothesized that metformin therapy will result in a higher ejection fraction after 4 months.
Time Frame: 4 months
Population: patients undergoing primary percutaneous coronary intervention (PCI) for STEMI
Measure: Mean (95% Confidence Interval); unit: % of LVEF
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 191 | 189
% of LVEF | 53.1 [51.6 to 54.6] | 54.8 [53.5 to 56.1]

2. Secondary Outcome: the Incidence of a Cardiovascular Event
Description: Cardiovascular events include major cardiac adverse events (MACE; death, recurrent MI, target lesion revascularization), stroke, non-elective hospitalizations for chest pain or heart failure, all recurrent coronary interventions, and internal cardiac defibrillator implantations. Mortality will be divided into cardiac and non-cardiac. Cardiac death will be divided into three categories: heart failure, sudden death and other. A cardiologist will confirm deaths from cardiovascular causes by examining medical records obtained from hospitals and attending physicians or from attending general practitioner if the patient died at home.
Time Frame: 4 months and longterm follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Markers of Heart Failure and Glycometabolic State
Description: markers of heart failure: neurohormones (e.g. NT-proBNP), renal function (e.g. MDRD); glycometabolic state: e.g. HbA1c.
Time Frame: 4 months and longterm follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Myocardial Infarct Size and Transmural Extent of Infarction as Measured With Cardiac Magnetic Resonance Imaging
Description: myocardial infarct size and transmural extent of infarction will be measured using Late Gadolinium Enhancement cardiac magnetic imaging
Time Frame: 4 months after hospitalization
Reporting Status: Not Posted

5. Secondary Outcome: Diastolic Function
Description: echocardiographic analysis of diastolic function
Time Frame: 4 months
Reporting Status: Not Posted

6. Secondary Outcome: Glycometabolic State
Description: measured by oral glucose tolerance testing and Glycated Hemoglobin according to current criteria
Time Frame: 4 months and long-term follow-up
Reporting Status: Not Posted

7. Secondary Outcome: Cardiac MRI After 4 Months, Per Protocol Analysis
Description: A per-protocol analysis, excluding patients diagnosed with new onset diabetes and treated with oral antihyperglycemic agents or insulin prior to cardiac MRI, will be performed as a secondary efficacy parameter
Time Frame: 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 3/191 | 1/188
Serious Adverse Events (participants affected / at risk) | 11/191 | 6/188
Other Adverse Events (participants affected / at risk) | 73/191 | 51/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=191) | Placebo (N=188)
Reinfarction (Cardiac disorders) | 8 (8) | 5 (5)
Cardiovascular death (Cardiac disorders) | 1 (1) | 0 (0)
Target lesion revascularization (Cardiac disorders) | 5 (5) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=191) | Placebo (N=188)
Non-target lesion revascularization (Cardiac disorders) | 40 (40) | 26 (26)
CABG (Cardiac disorders) | 10 (10) | 5 (5)
Hospitalization for chest pain (Cardiac disorders) | 23 (23) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes